CLINICAL TRIAL: NCT05566587
Title: Designing a Personalized Diet to Reduce the Risk of Crohn's Disease Onset
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Ken Croitoru, Clinician Scientist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: POP21-10037
Record Dates: First submitted 2022-09-16; First posted 2022-10-04 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Diet, Healthy; High Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western to Mediteranean to Western Diet (Other): Weeks 2 and 3 = WD Weeks 4 and 5 = MD Weeks 6 and 7 = WD
  Interventions: Other: Mediteranean to Western to Mediteranean Diet; Other: Western to Mediteranean to Western Diet
- Mediteranean to Western to Mediteranean Diet (Other): Weeks 2 and 3 = MD Weeks 4 and 5 = WD Weeks 6 and 7 = MD
  Interventions: Other: Mediteranean to Western to Mediteranean Diet; Other: Western to Mediteranean to Western Diet

INTERVENTIONS:
Other: Mediteranean to Western to Mediteranean Diet — week 2-3 : Switching between Mediterranean diet and Western diet week 4-5 : Switching between Western diet and Mediterranean diet week 6-7 : Switching between Mediterranean diet and Western diet
Other: Western to Mediteranean to Western Diet — week 2-3 : Switching between Western diet and Mediterranean diet week 4-5 : Switching between Mediterranean diet and Western diet week 6-7 : Switching between Western diet and Mediterranean diet

SUMMARY:
The purpose of this trial is to run a pilot study that examines the impact of different dietary components on risk factors such as the Genetic, Environmental, Microbial (GEM) Microbiome Risk Score (GMRS) and fecal calprotectin (FCP), a marker of inflammation in the bowels, and a risk factor for developing Crohn's disease (CD) among first degree relatives (parents, siblings, or offspring) of Crohn's patients. The study will utilize the Western diet and the Mediterranean diet to explore the complex interplay between diet, microbiome, and inflammatory biomarkers to identify specific dietary components that may be beneficial in reducing the risk of developing CD. The study will enroll 30 participants from Mount Sinai Hospital in Toronto.

DETAILED DESCRIPTION:
This study is a clinical trial that will occur at Mount Sinai Hospital and healthy first degree relatives of CD patients will be recruited. Participation will occur over 7 weeks with 1 week of consuming the subject's regular diet and 6 weeks of intervention. A total of 30 subjects are expected to be enrolled into this trial. As part of this trial, The study will attempt to modify dietary consumption between the Western Diet (WD) and the Mediterranean Diet (MD) to evaluate participants responses to specific food items key to the WD or MD by monitoring subject's GMRS and FCP. Subjects will be randomized into one of two groups (1:1), in which there will be crossover between the two diets. Stool samples will be collected 3 times a week, a daily questionnaire and a daily consumption diary will be completed through an app.

Group 1 will follow the WD for weeks 2 and 3, switch to the MD for weeks 4 and 5, and then back to the WD for weeks 6 and 7. Group 2 will follow the MD for weeks 2 and 3, switch to the WD for weeks 4 and 5, and then back to the MD for weeks 6 and 7.

Meal plans developed by the study Dietitian and recipes will be provided for all weeks of the intervention (weeks 2-7). These meal plans will be identical for subjects within the same group. Groceries required to prepare the meals as per the meal plan will be provided to subjects on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, asymptomatic first degree relative (child or sibling) of someone with Crohn's disease
* Have at least 1 bowel movement every other day

Exclusion Criteria:

* Received antibiotic treatment within 3 months of recruitment
* Unintentional weight loss in the last 3 months more than 15% of baseline weight
* Have ever been diagnosed with any chronic or recurring gastro-intestinal disease or bowel disease
* Belly pain occurred more than once per week for longer than three months in the past year
* Diarrhea (>three times per day) has been occurring for more than three months in the last year
* Have blood in their stool with most stools
* Diagnosed with diabetes
* Diagnosed with Celiac disease
* Diagnosed with irritable bowel syndrome
* Diagnosed with inflammatory bowel disease
* Presents significant symptoms of gastrointestinal disease
* Pregnant or breastfeeding women
* Has any serious food allergies
* Diagnosed with lactose intolerance
* Unable to stop NSAID or probiotic use during the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Personalized model | 7 weeks
  Repeated measures of FCP and GMRS will be used to generate a personalized model identifying food items that provide are predicted to have the greatest effect in the GMRS and FCP levels for a given individual

SECONDARY OUTCOMES:
Concentration of FCP levels over time during each intervention | Duration of each diet (2 to 4 weeks)
  fecal calprotectin will be analyzed from all stool samples collected during the study to provide continual data on any changes in intestinal inflammation
Modulation of GMRS over time during each intervention | Duration of each diet (2 to 4 weeks)
  Microbiome data will be collected from all stool samples collected during the study to provide continual data on any changes. This data will be used to calculate the GMRS at each time point. A higher GMRS indicate high risk for Crohn's disease
Measure of microbial taxa relative abundance over time during each intervention | Duration of each diet (2 to 4 weeks)
  Microbiome data will be collected from all stool samples collected during the study to provide continual data on any changes in microbial composition
Ability to maintain a balanced diet as measured by food intake records | 6 weeks
  Through the submission of the daily food diaries an assessment on the ability to maintain the diet will be reviewed
Adherence to the interventions | 6 weeks
  Compliance to the diet will be monitored through an app throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Croitoru, Principal Investigator — MOUNT SINAI HOSPITAL